CLINICAL TRIAL: NCT04567511
Title: Prospective, Single-Arm, Open-Label Use of Hemlibra (Emicizumab) in the Treatment of Mild Hemophilia A
Brief Title: Hemlibra in Mild Hemophilia A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana Hemophilia &Thrombosis Center, Inc. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Amy D Shapiro, MD, Medical Director, Indiana Hemophilia &Thrombosis Center, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RO-IIS-2019-20049
Record Dates: First submitted 2020-07-29; First posted 2020-09-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Factor VIII Deficiency, Congenital
Keywords: hemophilia A; mild hemophilia A; Factor VIII deficiency
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: single arm prospective open-label single-center study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients with mild hemophilia A (without inhibitors) will be treated with prophylactic emicizumab. The clinical hemostatic efficacy and safety will be assessed. Secondary outcomes will assess changes in quality of life and joint health in treated patients.
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — bispecific monoclonal antibody binding to activated Factor IX and Factor X
  Other Names: Hemlibra

SUMMARY:
This is a single arm, phase 4, prospective, open-label, United States single-center study to determine the hemostatic characteristics of Hemlibra (emicizumab) as measured by coagulation laboratory parameters in the mild hemophilia A male patient population with endogenous altered FVIII (baseline FVIII activity of >5% to 30%). The safety and hemostatic efficacy of Hemlibra (emicizumab) in this patient population will be investigated. Secondary outcomes will assess changes in joint health and quality of life in treated patients.

DETAILED DESCRIPTION:
This is a single arm, phase 4, prospective, open-label, United States single-center study to develop laboratory data and assess the clinical hemostatic efficacy and safety of Hemlibra (emicizumab) for hemostatic control of mild hemophilia A patients (baseline FVIII activity, >5 to 30%). Males aged ≥5 years to ≤45 years without inhibitors are eligible for enrollment. Secondary outcomes will assess changes in quality of life and joint health in treated patients.

Approximately 20 patients will be enrolled. As much as possible, the patient population will be selected to provide a variety of FVIII activity levels and F8 genetic defects.

Carrier females are not eligible for the study as the goal is to examine the effect of altered FVIII on Hemlibra (emicizumab) binding; carrier females with FVIII levels in the mild range of deficiency have one altered and one normal F8 gene that results in a mixture of both normal and altered FVIII proteins thereby complicating the interpretation of study results.

Patients with a FVIII inhibitor (or a history of a FVIII inhibitor) are not eligible for this study; if a subject develops a FVIII inhibitor during the study, they will be withdrawn from the study and offered the current standard of care.

Patients <5 years of age will be excluded from the study due to 1) the number of blood draws and the quantity of blood required; and 2) likelihood of reaching a minimum weight to utilize Stimate (~20 kg).

Patients with risk factors for thrombosis or TMA will be excluded from the study. Patients >45 years of age, >30 BMI, with a history of CVD, or >20% risk of CVD over a 10-year period using the atherosclerotic cardiovascular disease (ASCVD) risk estimator will also be excluded to minimize potential adverse events.

Patients with any number of FVIII exposure days are eligible for enrollment, as are previously untreated patients (PUPs). Although expected to be an uncommon occurrence, PUPs may be at risk of developing FVIII inhibitors while enrolled in the study due to exogenous FVIII exposure if required; as such they will be tested (bovine chromogenic modified inhibitor assay) after FVIII exposure per IHTC standard guidelines (after an episode of intensive treatment, between 3-5 EDs and then at 10 ED, etc.) Should a FVIII inhibitor develop in a PUP while on study, they will be removed from the study and offered the current standard of care.

To ensure no other bleeding disorders are present that might confound responses or lead to the development of a bleeding event unrelated to the underlying diagnosis of mild hemophilia A, a VWD panel and blood group will be obtained during screening.

Hemlibra (emicizumab) will be administered as weekly prophylaxis using the FDA-approved weekly dosing regimen following the enrollment/screening visit (first study visit) and the administration of the 4 weekly loading doses (second study visit). A choice of other approved dosing regimens (Q2W or Q4W) will not be offered as the primary regimen to limit variability in Cmin/Cmax exposure levels. The weekly prophylaxis regimen was selected to be the easiest for mild hemophilia A patients to remember as they are rarely on FVIII prophylaxis and infrequently need to administer on-demand hemostatic agents.

Bleeding events will be recorded and treated with locally available hemostatic agents (eg, Stimate [DDAVP/desmopressin acetate], pdFVIII, rFVIII, etc) as required. If FVIII is required for treatment of a bleeding event, the dose expected to achieve hemostasis will be utilized.

The enrollment period is 37 months; with a total study period of 60 months. The study comprises 2 parts following screening. Subjects will initially be enrolled in Part A (12 months) including a 1-month period of Hemlibra dose administration and collection of baseline laboratory data, with the option of enrolling in part B (12 months) upon successful completion of Part A and approval of the Study Investigator. Up to a 1-month window is provided between screening and administration of the first loading dose, depending on the return of required laboratory testing data and subject availability. When subjects complete the study, they will be requested to meet with their IHTC hemophilia physician to resume their previous therapeutic regimen or be offered the current standard of care.

Part A Loading dose administration (month 1 ±2 days):

This is a 1-month (±2 days) period during which the 4 weekly loading doses of Hemlibra (emicizumab) will be administered. Additionally, baseline laboratory data, banked plasma samples, MSKUS imaging and quality of life questionnaires will be completed.

Part A Maintenance Hemlibra therapy [months 2-13 (±2 weeks)]:

The purpose of this section of Part A is to collect laboratory data to determine the impact of Hemlibra (emicizumab) on laboratory coagulation parameters including thrombin generation in patients with circulating levels of endogenous altered FVIII (>5% to 30% baseline FVIII activity). Laboratory data will be collected at month 4 (±2 weeks), month 7 (±2 weeks) and month 13 (±2 weeks). Additional data, including bleeding events, bleed treatment, intercurrent procedures, quality of life (Haemo-QoL and CATCH questionnaires if <17 years of age; Haem-A-QoL and CATCH questionnaires if ≥17 years of age) and joint health (MSKUS) will be collected at baseline and 12 months (±2 weeks).

A Stimate/DDAVP challenge may occur at either the 4-month (±2 weeks) or 7-month (±2 weeks) study visit to investigate the hemostatic characteristics of Hemlibra (emicizumab) in the presence of elevated levels of altered FVIII using coagulation laboratory assays. The Stimate/DDAVP challenge will not be performed if the patient has a documented history of lack of response as defined by an increase of FVIII < 2 times baseline level. The Stimate/DDAVP challenge may be delayed to a later study visit due to recent treatment (within the previous 4 days) with a FVIII concentrate or Stimate (DDAVP/desmopressin acetate) or for convenience (at the discretion of the Study Investigator). The Stimate/DDAVP challenge may also be delayed or its route of administration altered if a subject weighs ≥10kg to <20kg; a weight-based subcutaneous dose of DDAVP/desmopressin acetate may be administered for subjects <20 kg at the discretion of the Study Investigator). The Stimate/DDAVP challenge may be delayed to a later study visit if the intranasal route of administration is compromised and subcutaneous administration of DDAVP/desmopressin acetate is not planned. See Section 3.1.9 for full details on the Stimate/DDAVP challenge.

Part B [months 14-25 (±2 weeks)]:

Upon successful completion of Part A, subjects may continue Hemlibra (emicizumab) treatment by enrolling in Part B if approved by the Study Investigator and per patient desire to continue treatment. The goal of Part B is to acquire additional data on bleeding events, bleed treatment, intercurrent procedures, changes in quality of life (Haemo-QoL and CATCH questionnaires if <17 years of age; Haem-A-QoL and CATCH questionnaires if ≥17 years of age) and joint health (MSKUS). This extended collection period is desired due to the infrequent and variable ABR in individuals with mild hemophilia A. Subjects will receive Hemlibra (emicizumab treatment in Part B for 12 months.

The study is seeking to address the following knowledge gaps:

* Is Hemlibra (emicizumab)-conferred hemostatic coverage additive to the activity of the endogenous altered FVIII protein in mild hemophilia A patients or is there evidence that endogenous altered FVIII protein is competitive with Hemlibra (emicizumab)?
* Do specific FVIII mutations confer more or less additive or competitive effect? In silico simulations of the altered protein (based upon the patient's genetic alteration) may be investigated to predict the protein's in vivo function and interaction with Hemlibra (emicizumab) binding (secondary exploratory goal)
* What is the hemostatic contribution of Hemlibra (emicizumab) in the presence of maximal endogenous altered FVIII protein release (Stimate/DDAVP challenge with coagulation laboratory assays)?
* Are there patients with specific genetic mutations who would benefit from Hemlibra (emicizumab) usage, or can a sub-population of patients of mild hemophilia be identified for whom Hemlibra (emicizumab) would not represent optimal therapy?
* Is weekly Hemlibra (emicizumab) safe to administer in patients with mild hemophilia A and does it reduce the incidence of bleeding events or the need for alternate hemostatic agents, including during/following surgeries and procedures?
* Does weekly prophylactic Hemlibra (emicizumab) result in an increase in QoL and/or activity in mild hemophilia A patients?
* Does weekly prophylactic Hemlibra (emicizumab) result in an improvement in joint health (ie, the control of progression, stabilization or regression of joint damage) using 6 joint point of care musculoskeletal

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form from the subject, parent or guardian
* Male sex
* Diagnosis of mild congenital hemophilia A (baseline FVIII level of >5% to 30%) without a current FVIII inhibitor or a history of FVIII inhibitor
* Any number of FVIII exposure days, including PUPs
* BMI <30
* Age ≥5 years to ≤45 years
* Medical documentation of bleeding events, outcomes and hemostatic product usage for 12 months prior to study enrollment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including the health-related questionnaires, activity tracking, and bleed diaries, using systems provided during the study
* Willingness to undergo a Stimate/DDAVP challenge (only if the subject reports no adverse event associated with prior Stimate [DDAVP/desmopressin acetate] use); Stimate/DDAVP challenge will not be performed if the patient has a documented history of lack of response as defined by an increase of FVIII < 2 times baseline level
* Adequate hepatic function, defined as total bilirubin ≤1.5 × age-adapted upper limit of normal (ULN) (excluding Gilbert's syndrome) and both AST and ALT ≤3 × age-adapted ULN at the time of screening, and no clinical signs or known laboratory/radiographic evidence consistent with cirrhosis
* Adequate hematologic function, defined as a platelet count ≥100,000/μL and a PT≤1.5 times the ULN at the time of screening
* Adequate renal function, defined as serum creatinine ≤2.5 × age-adapted ULN and creatinine clearance ≥30 mL/min by Cockcroft-Gault formula

Exclusion Criteria:

* Inherited or acquired bleeding disorder other than mild congenital hemophilia A (baseline FVIII level of >5% to 30%)
* Any bleeding disorder other than or in addition to mild hemophilia A
* Current or prior inhibitor to FVIII (any titer)
* Female sex
* History of CVD, risk of CVD by the ASCVD risk estimator (defined as a subject having >20% risk of a cardiovascular event within the next 10 years if the subject is ≥20 years of age) and/or a history of ischemic heart disease [ICD codes 120-125]
* High risk for TMA (eg, have a previous medical or family history of TMA), in the Study Investigator's judgment
* History of illicit drug or alcohol abuse by report or in the Study Investigator's judgment
* Previous (within the last 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* Other conditions (eg, certain autoimmune diseases) that may currently increase the risk of bleeding or thrombosis
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the Hemlibra (emicizumab) injection
* Known HIV infection with CD4 counts <200 cells/μL. HIV infection with CD4 counts ≥200 cells/μL permitted
* Use of systemic immunomodulators (eg, interferon) at enrollment or planned use during the study, with the exception of anti-retroviral therapy
* Concomitant disease, condition, significant abnormality on screening evaluations or laboratory tests, or treatment that could interfere with the conduct of the study, or that would, in the opinion of the Study Investigator, pose an additional unacceptable risk in administering study drug to the patient
* Receipt of any of the following:

  * Hemlibra (emicizumab) in a prior investigational study
  * An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration
  * A non-hemophilia-related investigational drug within last 30 days or 5 half-lives, whichever is shorter
  * Any other investigational drug currently being administered or planned to be administered
* Inability to comply with the study protocol in the opinion of the Study Investigator

Ages: 5 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — only males will be enrolled in the study.
Enrollment: 20 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Interaction of Hemlibra (emicizumab) binding with endogenous altered FVIII protein in an individual with mild hemophilia A and the combined effect on thrombin generation and hemostatic characteristics | Before treatment, month 4, month 7, and month 13
  Change in FVIII human chromogenic activity, FVIII bovine chromogenic activity, and Thrombin Generation Assay relatively to one another

SECONDARY OUTCOMES:
Breakthrough bleeds | Through study completion, up to 35 months
  Rate of bleeding events requiring alternate hemostatic therapy
Factor VIII alteration and coagulation | Before treatment, month 4, month 7, and month 13
  Relationship between Factor VIII alteration and coagulation laboratory parameters
Change from baseline joint disease annually | Through study completion annually, up to 35 months
  Baseline presence of joint disease through 6 joint POC MSKUS and its stabilization, resolution, or progression
AE, SAE, and ADA | Through study completion annually, up to 35 months
  Rate of adverse events (AEs) and serious adverse events (SAEs) including lack of efficacy and development of neutralizing anti-drug antibodies (ADA)
ADA development | ADA assay at month 4, month 7, month 13, and end of study participation
  Number of participants with development of neutralizing anti-drug antibodies (ADA) if it occurs
Alternate hemostatic therapies with surgery | At time of patient's surgery if applicable
  Rate of use of alternate hemostatic therapies (eg, FVIII, Stimate/DDAVP, etc) during surgeries and procedures and their hemostatic efficacy to prevent or treat bleeding
Change in quality of life: questionnaire | Before treatment, Day 0, Day 7, Day 14, Day 21, month 13, month 25
  Change in quality of life as measured by Haemo-QoL (haemophilia-specific quality of life questionnaire) if <17 years of age; and Haem-A-QoL-A (haemophilia-specific quality of life questionnaire for adults) if ≥17 years of age. Scores range from 0 to 100, with higher scores indicating a lower quality of life.
Change in activity: questionnaire | Before treatment, Day 0, Day 7, Day 14, Day 21, month 13, month 25
  Change in activity level as measured by CATCH (Comprehensive Assessment Tool of Challenges in Hemophilia) questionnaire. Change from baseline in the daily activity risk perception and impact domain score over time. This is not a scaled assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Shapiro, MD, Principal Investigator — Indiana Hemophilia &Thrombosis Center, Inc.
Locations (1):
- Indiana Hemophila @Thrombosis Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share resources and data from this project through collaborative publications in the scientific literature as well as through national, regional and international conference presentations. The investigators will also share our methods and findings in a prompt manner with regional, national and international stakeholders to ensure that findings will be readily available to other researchers and clinicians with clinical or scientific interest in the subject area. Individual participant data that underlie the results reports in publications, reports or presentations (including text, tables, figures and appendices) will be shared after de-identification.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and additional information on study methods will be made available starting 9 months after publication or conclusion of the study and ending 36 months following publication or study conclusion.
Access Criteria: IPD and study information will be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary"), whose proposals are methodologically sound, and for purposes that are consistent with the aims of the underlying research. Proposals will be reviewed by the Principle Investigator, Dr. Amy Shapiro, and may be submitted to ashapiro@ihtc.org. Requestors will be required to sign a data access and use agreement.

REFERENCES:
- [Result] Batorova A, Holme P, Gringeri A, Richards M, Hermans C, Altisent C, Lopez-Fernandez M, Fijnvandraat K; European Haemophilia Treatment Standardisation Board. Continuous infusion in haemophilia: current practice in Europe. Haemophilia. 2012 Sep;18(5):753-9. doi: 10.1111/j.1365-2516.2012.02810.x. Epub 2012 Apr 25. PMID 22530687
- [Result] Blanchette VS, Key NS, Ljung LR, Manco-Johnson MJ, van den Berg HM, Srivastava A; Subcommittee on Factor VIII, Factor IX and Rare Coagulation Disorders of the Scientific and Standardization Committee of the International Society on Thrombosis and Hemostasis. Definitions in hemophilia: communication from the SSC of the ISTH. J Thromb Haemost. 2014 Nov;12(11):1935-9. doi: 10.1111/jth.12672. Epub 2014 Sep 3. No abstract available. PMID 25059285
- [Result] Centers for Disease Control and Prevention (2014). Hemophilia Data & Statistics Retrieved April 22, 2014, from http://www.cdc.gov/ncbddd/hemophilia/data.html
- [Result] Franchini M, Favaloro EJ, Lippi G. Mild hemophilia A. J Thromb Haemost. 2010 Mar;8(3):421-32. doi: 10.1111/j.1538-7836.2009.03717.x. Epub 2009 Dec 7. PMID 19995408
- [Result] Franchini M, Mannucci PM. Hemophilia A in the third millennium. Blood Rev. 2013 Jul;27(4):179-84. doi: 10.1016/j.blre.2013.06.002. Epub 2013 Jun 28. PMID 23815950
- [Result] Franchini M, Mannucci PM. Inhibitor eradication with rituximab in haemophilia: where do we stand? Br J Haematol. 2014 Jun;165(5):600-8. doi: 10.1111/bjh.12829. Epub 2014 Mar 15. PMID 24628543
- [Result] Gringeri A, Leissinger C, Cortesi PA, Jo H, Fusco F, Riva S, Antmen B, Berntorp E, Biasoli C, Carpenter S, Kavakli K, Morfini M, Negrier C, Rocino A, Schramm W, Windyga J, Zulfikar B, Mantovani LG. Health-related quality of life in patients with haemophilia and inhibitors on prophylaxis with anti-inhibitor complex concentrate: results from the Pro-FEIBA study. Haemophilia. 2013 Sep;19(5):736-43. doi: 10.1111/hae.12178. Epub 2013 Jun 4. PMID 23731246
- [Result] Hay CR. Factor VIII inhibitors in mild and moderate-severity haemophilia A. Haemophilia. 1998 Jul;4(4):558-63. doi: 10.1046/j.1365-2516.1998.440558.x. PMID 9873794
- [Result] Kempton CL, Allen G, Hord J, Kruse-Jarres R, Pruthi RK, Walsh C, Young G, Soucie JM. Eradication of factor VIII inhibitors in patients with mild and moderate hemophilia A. Am J Hematol. 2012 Sep;87(9):933-6. doi: 10.1002/ajh.23269. Epub 2012 Jun 26. PMID 22733686
- [Result] Mahlangu J, Oldenburg J, Paz-Priel I, Negrier C, Niggli M, Mancuso ME, Schmitt C, Jimenez-Yuste V, Kempton C, Dhalluin C, Callaghan MU, Bujan W, Shima M, Adamkewicz JI, Asikanius E, Levy GG, Kruse-Jarres R. Emicizumab Prophylaxis in Patients Who Have Hemophilia A without Inhibitors. N Engl J Med. 2018 Aug 30;379(9):811-822. doi: 10.1056/NEJMoa1803550. PMID 30157389
- [Result] Makris M, Oldenburg J, Mauser-Bunschoten EP, Peerlinck K, Castaman G, Fijnvandraat K; subcommittee on Factor VIII, Factor IX and Rare Bleeding Disorders. The definition, diagnosis and management of mild hemophilia A: communication from the SSC of the ISTH. J Thromb Haemost. 2018 Dec;16(12):2530-2533. doi: 10.1111/jth.14315. Epub 2018 Nov 15. No abstract available. PMID 30430726
- [Result] National Institutes of Health (2014). What Is Hemophilia? Retrieved April 22, 2014, from https://www.nhlbi.nih.gov/health/health-topics/topics/hemophilia/
- [Result] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557
- [Result] Pezeshkpoor B, Gazorpak M, Berkemeier AC, Singer H, Pavlova A, Biswas A, Oldenburg J. In silico and in vitro evaluation of the impact of mutations in non-severe haemophilia A patients on assay discrepancies. Ann Hematol. 2019 Aug;98(8):1855-1865. doi: 10.1007/s00277-019-03691-1. Epub 2019 Apr 17. PMID 30997536
- [Result] Pipe, S. (2018). Emicizumab subcutaneous dosing every 4 weeks is safe and efficacious in the control of bleeding in persons with haemophilia A with and without inhibitors - Results from the phase 3 HAVEN 4 study. World Federation of Hemophila World Congress Glasgow, Scotland.
- [Result] Prelog T, Dolnicar MB, Kitanovski L. Low-dose continuous infusion of factor VIII in patients with haemophilia A. Blood Transfus. 2016 Sep;14(5):474-80. doi: 10.2450/2015.0080-15. Epub 2015 Nov 16. PMID 26674820
- [Result] Sengupta M, Sarkar D, Ganguly K, Sengupta D, Bhaskar S, Ray K. In silico analyses of missense mutations in coagulation factor VIII: identification of severity determinants of haemophilia A. Haemophilia. 2015 Sep;21(5):662-9. doi: 10.1111/hae.12662. Epub 2015 Apr 9. PMID 25854144
- [Result] Shima, M., K. Nogami, S. Nagami, S. Yoshida, K. Yoneyama, A. Ishiguro, T. Suzuki and M. Taki (2018) Every 2 Weeks or Every 4 Weeks Subcutaneous Injection of Emicizumab in Pediatric Patients with Severe Hemophilia A without Inhibitors: A Multi-Center, Open-Label Study in Japan (HOHOEMI Study). Blood 132:1186-1186.
- [Result] World Federation of Hemophilia (2012). Guidelines for the management of hemophilia Retrieved February 16, 2015, from http://www1.wfh.org/publication/files/pdf-1472.pdf
- [Result] World Federation of Hemophilia (2012). World Federation of Hemophilia report on the annual global survey 2011 Retrieved December 20, 2016, from http://www1.wfh.org/publication/files/pdf-1488.pdf
- [Result] World Federation of Hemophilia (2013). World Federation of Hemophilia report on the annual global survey 2013 Retrieved February 5, 2015, from http://www1.wfh.org/publications/files/pdf-1591.pdf
- [Result] World Federation of Hemophilia (2016). World Federation of Hemophilia report on the annual global survey 2015 Retrieved December 20, 2016, from http://www1.wfh.org/publication/files/pdf-1669.pdf.
- [Result] World Federation of Hemophilia (2017). World Federation of Hemophilia Annual Global Survey Data Retrieved May 30, 2017, from https://www.wfh.org/en/resources/annual-global-survey
- [Result] Young G, Liesner R, Chang T, Sidonio R, Oldenburg J, Jimenez-Yuste V, Mahlangu J, Kruse-Jarres R, Wang M, Uguen M, Doral MY, Wright LY, Schmitt C, Levy GG, Shima M, Mancuso ME. A multicenter, open-label phase 3 study of emicizumab prophylaxis in children with hemophilia A with inhibitors. Blood. 2019 Dec 12;134(24):2127-2138. doi: 10.1182/blood.2019001869. PMID 31697801